CLINICAL TRIAL: NCT04176406
Title: Using fMRI-guided TMS to Increase Central Executive Function in Older Adults (MCI_Sub)
Acronym: MCI_Sub
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19, Funding ended
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00065334_1
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- rTMS over a node within the fronto-parietal network (Active Comparator): excitatory 5Hz rTMS will be applied over a node within the fronto-parietal network, defined via network analysis.
  Interventions: Device: rTMS
- Sham rTMS over a node within the fronto-parietal network (Sham Comparator): electrical sham coil applied over a node within the fronto-parietal network.
  Interventions: Device: Sham rTMS
- rTMS over the DLPFC (Active Comparator): excitatory 5Hz rTMS will be applied over the dorso-lateral prefrontal cortex showing the strongest fMRI activation.
  Interventions: Device: rTMS
- Sham rTMS over the DLPFC (Sham Comparator): electrical sham coil applied over the DLPFC.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — excitatory 5Hz rTMS will be used
  Arms: rTMS over a node within the fronto-parietal network; rTMS over the DLPFC
Device: Sham rTMS — an electrical sham coil reproducing the same clicking sound and tactile sensation than the active rTMS will be used
  Arms: Sham rTMS over a node within the fronto-parietal network; Sham rTMS over the DLPFC

SUMMARY:
This is an administrative supplement to an existing project "Using fMRI-guided TMS to increase central executive function in older adults: NCT02767323" This award allows extending our existing fMRI-TMS paradigm to patients with a prodromal form of Alzheimer's Disease (AD) known as amnestic Mild Cognitive Impairment (MCI), and investigate the role of brain health factors in mediating the TMS-related memory performance benefits associated with communication between a network of frontoparietal brain regions in these populations.

The focus on focal neurostimulation at only a single site represents a fundamental gap in the approach of memory-based neurostimulation therapies. Neurostimulation affects multiple sites within a cortical network, but these global effects have not been used as targets for stimulation because of limited knowledge about what influence these localized sites have on global changes in brain state. To address this problem, multimodal neuroimaging tools and network modeling approaches developed though the parent U01 project will be used, to demonstrate how focal neurostimulation improves the efficacy of TMS for enhancing memory function. These goals will be addressed in the Administrative Supplement under our two specific aims. First, network-guided TMS will be applied to optimize memory success based in the frontoparietal network (FPN) in a new group of MCI patients. A new form of TMS targeting that involves modeling of the global network to understand how the controllability of a stimulation site evokes changes in widespread brain networks will be tested. Second, structural and functional factors affecting the efficacy of individualized network-guided TMS will be identified to ameliorate deficits in MCI. By creating a multimodal model of neural deficits related to MCI, network-guided TMS will be adjusted to demonstrate how the MCI brain might compensate for these neural deficits. The parent U01 project has made foundational advances towards these goals, as we have demonstrated the ability of to selectively enhance and reduce working memory performance in healthy older adults. In the current Administrative Supplement this paradigm will be extended to a group of MCI participants in order to test the hypothesis that excitatory rTMS to the working memory network can provide positive outcomes for patients with pre-clinical AD. The proposed work will provide an important tool for studying the stability and controllability of network connectivity of memory states in the aging brain, as well as new information on the effectiveness of brain stimulation technologies as a therapeutic approach for cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* willing to provide consent
* signed HIPAA authorization
* clinical consensus for MCI; and/or met inclusion criterial on MoCA, ApoE.

Exclusion Criteria:

* History of any I DSM IV disorder that is unstable or untreated
* current or past history of substance abuse or dependence (excluding nicotine)
* women who are pregnant or breast feeding
* intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes
* increased risk of seizure for any reason, including prior diagnosis of epilepsy, seizure disorder, increased intracranial pressure, or history of significant head trauma greater than mild concussion (History of significant head trauma, including with loss of consciousness for ≥ 30 minutes, alteration of consciousness for up to 24 hours following the event, or post-traumatic amnesia) in the past 10yrs or head injury received after age 65
* Neurological disorder including, but not limited to: space occupying brain lesion; any history of seizures, history of cerebrovascular accident; cerebral aneurysm , Dementia, Huntington chorea, multiple sclerosis
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that are on the strong potential hazard list for rTMS.
* Subjects taking medications with an ACB score of 3.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence G Appelbaum, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated prior to application of rTMS or Sham.
Period: Overall Study
Arm/Group | rTMS Over a Node Within the Fronto-parietal Network | Sham rTMS Over a Node Within the Fronto-parietal Network | rTMS Over the DLPFC | Sham rTMS Over the DLPFC
Started (None of the participants were randomized to any of the Arms/Groups) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: These participants only performed the behavioral task. No TMS was applied.
Groups:
- Enrolled Participants: The following numbers represent the baseline characteristics for the participants enrolled in the study, who performed only the behavioral task. None of these participants received rTMS
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Acute Effect of a rTMS Session on the Performance for a Working Memory Task, as Measured by Accuracy (in Percentage)
Description: Accuracy (in percentage) will be assessed to evaluate the acute effect of rTMS.
Time Frame: Through study completion, an average of one year
Population: The study had to be interrupted because of Covid-19 situation, while we were still piloting the behavioral task. Therefore no data with rTMS were collected.
Arm/Group | Sham rTMS Over the DLPFC
Number analyzed (Participants) | 0

2. Primary Outcome: Acute Effect of a rTMS Session on the Performance for a Working Memory Task, as Measured by Reaction Times (ms)
Description: Reaction times (in ms) will be assessed to evaluate the acute effect of rTMS
Time Frame: Through study completion an average of one year
Population: The study had be be terminated early due to the Covid-19 situation, while we were still piloting the behavioral task. Therefore no participants received rTMS
Arm/Group | rTMS Over a Node Within the Fronto-parietal Network | Sham rTMS Over a Node Within the Fronto-parietal Network | rTMS Over the DLPFC | Sham rTMS Over the DLPFC
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: adverse event data are collected during rTMS and a few minutes after.
Description: rTMS was not applied so no adverse event/ all cause mortality were monitored
Arm/Group | rTMS Over a Node Within the Fronto-parietal Network | Sham rTMS Over a Node Within the Fronto-parietal Network | rTMS Over the DLPFC | Sham rTMS Over the DLPFC
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT04176406/Prot_SAP_000.pdf